CLINICAL TRIAL: NCT06421129
Title: Identifying Landmark Factors of Anal Fistulas Through Predictive Modeling for Adverse Surgical Outcomes: a Retrospective Cohort Study
Brief Title: Identifying Landmark Factors of Anal Fistulas
Status: Completed | Type: Observational
Sponsor: Guanlin Liu (Other)
Responsible Party: Sponsor-Investigator, Guanlin Liu, Principal Investigator, First Hospital of China Medical University
Organization: First Hospital of China Medical University (Other)
Other Study IDs: Number: 2024【546】
Record Dates: First submitted 2024-05-10; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Anal Fistulas; Anal Fistula
Keywords: anal fistula; perianal and rectal spaces; surgery
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- good prognosis: A good prognosis within 1-year post-surgery was defined as healing of the internal and external openings of the fistula, no recurrence of the fistula, no secondary perianal infection, no symptoms of incontinence, no persistent pain, and the ability of the patient to perform activities independently
  Interventions: Procedure: anal fistula surgery
- poor prognosis: outcomes that did not meet good prognosis criteria indicated a poor prognosis
  Interventions: Procedure: anal fistula surgery

INTERVENTIONS:
Procedure: anal fistula surgery — anal fistula surgery consists of;Fistulotomy and Fistulotomy with seton placement

SUMMARY:
The goal of this observational study is to understand the effects of anatomical factors, etiology, and complexity of anal fistula on the prognosis of patients undergoing anal fistula surgery within one year post-operation.The main question it aims to answer is:

Which factors are indicative of the prognosis of anal fistula surgery? Which factors are landmark factors of anal fistulas?

Participants who have already undergone anal fistula surgery at our hospital will receive outpatient and telephone follow-up to assess their prognosis.

DETAILED DESCRIPTION:
The search function of the electronic medical record system and surgical records were used to screen patients. For the enrolled patients, the electronic medical record system, imaging report query system, medical order system, outpatient follow-up and telephone follow-up were used to collect data Data were entered into Excel 2021 (Microsoft Corp., Redmond, WA, USA) and checked for errors before conducting statistical analyses using R software (version 4.2.2; The R Foundation, Vienna, Austria).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with an anal fistula through clinical and radiological examinations; surgeries performed by physicians at our hospital who had at least a title of Associate Chief Physician, with operative records completed after surgery; patients with complete clinical data; and patients who completed post-operative outpatient follow-up and agreed to participate in telephone follow-up surveys.

Exclusion Criteria:

* Patients who were assessed clinically as unable to tolerate surgery; patients who refused surgical treatment; and patients who failed to complete the outpatient follow-up, refused telephone follow-up, or were lost to follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective cohort study was conducted at The First Affiliated Hospital of China Medical University
Sampling Method: Non-Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
history of perianal abscess and fistula | between 1 January 2020 and 1 February 2023
  Electronic medical record collection
Age | between 1 January 2020 and 1 February 2023
  Electronic medical record collection
History of underlying diseases | between 1 January 2020 and 1 February 2023
  Hypertension, heart disease and diabetes (Electronic medical record collection)
perianal and perirectal space involvement-perianal subcutaneous space | between 1 January 2020 and 1 February 2023
  Preoperative imaging examination data, electronic medical and record-surgery records were collected. The extent of anal fistula invasion into the perianal and rectal spaces was assessed based on preoperative imaging examinations and observations made during surgery. All surgical procedures were performed and documented by Associate Chief Physicians in our department. In cases in which the intraoperative findings differed from the imaging results, the findings observed during surgery were considered definitive.
perianal and perirectal space involvement-Posterior superficial anal space | between 1 January 2020 and 1 February 2023
  Preoperative imaging examination data, electronic medical and record-surgery records were collected. The extent of anal fistula invasion into the perianal and rectal spaces was assessed based on preoperative imaging examinations and observations made during surgery. All surgical procedures were performed and documented by Associate Chief Physicians in our department. In cases in which the intraoperative findings differed from the imaging results, the findings observed during surgery were considered definitive.
perianal and perirectal space involvement-Deep posterior anal space | between 1 January 2020 and 1 February 2023
  Preoperative imaging examination data, electronic medical and record-surgery records were collected. The extent of anal fistula invasion into the perianal and rectal spaces was assessed based on preoperative imaging examinations and observations made during surgery. All surgical procedures were performed and documented by Associate Chief Physicians in our department. In cases in which the intraoperative findings differed from the imaging results, the findings observed during surgery were considered definitive.
perianal and perirectal space involvement-Anterior superficial anal space | between 1 January 2020 and 1 February 2023
  Preoperative imaging examination data, electronic medical and record-surgery records were collected. The extent of anal fistula invasion into the perianal and rectal spaces was assessed based on preoperative imaging examinations and observations made during surgery. All surgical procedures were performed and documented by Associate Chief Physicians in our department. In cases in which the intraoperative findings differed from the imaging results, the findings observed during surgery were considered definitive.
perianal and perirectal space involvement-Deep anterior anal space | between 1 January 2020 and 1 February 2023
  Preoperative imaging examination data, electronic medical and record-surgery records were collected. The extent of anal fistula invasion into the perianal and rectal spaces was assessed based on preoperative imaging examinations and observations made during surgery. All surgical procedures were performed and documented by Associate Chief Physicians in our department. In cases in which the intraoperative findings differed from the imaging results, the findings observed during surgery were considered definitive.
perianal and perirectal space involvement-Submucosal space | between 1 January 2020 and 1 February 2023
  Preoperative imaging examination data, electronic medical and record-surgery records were collected. The extent of anal fistula invasion into the perianal and rectal spaces was assessed based on preoperative imaging examinations and observations made during surgery. All surgical procedures were performed and documented by Associate Chief Physicians in our department. In cases in which the intraoperative findings differed from the imaging results, the findings observed during surgery were considered definitive.
perianal and perirectal space involvement-Intersphincteric anal space | between 1 January 2020 and 1 February 2023
  Preoperative imaging examination data, electronic medical and record-surgery records were collected. The extent of anal fistula invasion into the perianal and rectal spaces was assessed based on preoperative imaging examinations and observations made during surgery. All surgical procedures were performed and documented by Associate Chief Physicians in our department. In cases in which the intraoperative findings differed from the imaging results, the findings observed during surgery were considered definitive.
Fistula origin | between 1 January 2020 and 1 February 2023
  Electronic medical record collection
fistula traversal through the internal and external sphincters | between 1 January 2020 and 1 February 2023
  Preoperative imaging examination data, electronic medical and record-surgery records were collected. The extent of anal fistula invasion into the anal sphincters was assessed based on preoperative imaging examinations and observations made during surgery. All surgical procedures were performed and documented by Associate Chief Physicians in our department. In cases in which the intraoperative findings differed from the imaging results, the findings observed during surgery were considered definitive.
perianal and perirectal space involvement-Ischioanal space | between 1 January 2020 and 1 February 2023
  Preoperative imaging examination data, electronic medical and record-surgery records were collected.The extent of anal fistula invasion into the perianal and rectal spaces was assessed based on preoperative imaging examinations and observations made during surgery. All surgical procedures were performed and documented by Associate Chief Physicians in our department. In cases in which the intraoperative findings differed from the imaging results, the findings observed during surgery were considered definitive.
perianal and perirectal space involvement-Ischiorectal space | between 1 January 2020 and 1 February 2023
  Preoperative imaging examination data, electronic medical and record-surgery records were collected. The extent of anal fistula invasion into the perianal and rectal spaces was assessed based on preoperative imaging examinations and observations made during surgery. All surgical procedures were performed and documented by Associate Chief Physicians in our department. In cases in which the intraoperative findings differed from the imaging results, the findings observed during surgery were considered definitive.
perianal and perirectal space involvement-Pelvirectal space | between 1 January 2020 and 1 February 2023
  Preoperative imaging examination data, electronic medical and record-surgery records were collected. The extent of anal fistula invasion into the perianal and rectal spaces was assessed based on preoperative imaging examinations and observations made during surgery. All surgical procedures were performed and documented by Associate Chief Physicians in our department. In cases in which the intraoperative findings differed from the imaging results, the findings observed during surgery were considered definitive.

SECONDARY OUTCOMES:
Sex | between 1 January 2020 and 1 February 2023
  Electronic medical record collection
Duration of preoperative symptoms | between 1 January 2020 and 1 February 2023
  Electronic medical record collection
Smoking history | between 1 January 2020 and 1 February 2023
  Electronic medical record collection
Anesthesia method | between 1 January 2020 and 1 February 2023
  Electronic medical record collection
Alcohol history | between 1 January 2020 and 1 February 2023
  Electronic medical record collection

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Meng, Study Director — First Hospital of China Medical University
Locations (1):
- The First Affiliated Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Six months after the completion of the experiment
Access Criteria: This study contains clinical data from medical records in our hospital. The datasets used and/or analysed during the current study are available from the study leader on reasonable request.
URL: https://clinicaltrials.gov